CLINICAL TRIAL: NCT07108062
Title: Using Tele-rehabilitation on Management of Pediatric Nocturnal Enuresis: Randomized Controlled Trial
Brief Title: Using Tele-rehabilitation on Management of Pediatric Nocturnal Enuresis
Acronym: UTMPNE
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hungarian University of Sports Science (Other)
Collaborators: Kafrelsheikh University (Other)
Responsible Party: Principal Investigator, Mohamed Abdelaziz Emam, Lecturer assistant at of Basic Sciences Department , Faculty of Physical Therapy, Kafrelsheikh Univerisity, Kafrelsheikh 33511, Egypt | PhD Researcher Hungarian University of Sports science, Budapest, Hungary, Kafrelsheikh University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KFSIRB200-671
Record Dates: First submitted 2025-07-29; First posted 2025-08-06 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-07

CONDITIONS: Enuresis Nocturnal; Urinary Incontinence
Keywords: Enuresis; Bedwetting; Urinary Incontinence; Nocturnal
MeSH Terms: conditions — Nocturnal Enuresis; Urinary Incontinence; Enuresis

STUDY DESIGN:
Intervention Model Description: participants are randomly assigned to one of two groups, and each group receives a different intervention
  Study Group: Receives telerehabilitation (lifestyle + dietary advice)
  Control Group: Does not receive telerehabilitation
  Participants in each group are treated simultaneously but independently, which is the hallmark of a parallel design.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study Group (Experimental): Receives Tele-rehabilitation (lifestyle + dietary advice)
  Interventions: Other: Experimental
- Control Group (Placebo Comparator): Does not receive tele-rehabilitation
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Experimental — (lifestyle + dietary advice)
  Arms: Study Group
Other: Placebo — No intervention
  Arms: Control Group

SUMMARY:
Objective:

To evaluate the effectiveness of telerehabilitation (via lifestyle and dietary advice) in managing primary nocturnal enuresis (bedwetting) in children aged 5-10 years.

Background:

Nocturnal enuresis is common in children and can be influenced by genetic, hormonal, and bladder-related factors. Treatment includes behavioral, pharmacological, and psychological approaches. Telerehabilitation-remote delivery of care-emerged during the COVID-19 pandemic as a promising tool for maintaining continuity of care.

Methodology:

Design: Randomized Controlled Trial

Participants: Children aged 5-10 with primary NE (wetting ≥4 nights/week), recruited online.

Exclusion: Children with secondary NE due to medical conditions or those on medication.

Groups:

Study group: Received telerehabilitation (lifestyle + dietary guidance).

Control group: No telerehabilitation.

Duration: 3 weeks (1 week baseline, 1 week intervention, 1 week follow-up)

Assessment:

Number of wet nights per week (using ICCS classification: responders, partial responders, non-responders)

Pediatric quality of life

Intervention Details:

Telerehabilitation involved dietary recommendations (e.g., reducing evening fluid intake, avoiding caffeine/chocolate), lifestyle tips, and motivational counseling delivered remotely to caregivers.

Data Analysis:

Pre- and post-intervention outcomes compared using paired t-tests. Demographics and clinical characteristics recorded.

DETAILED DESCRIPTION:
Introduction & Background:

Nocturnal Enuresis (NE) is the involuntary urination during sleep in children over 5 years of age, commonly known as bedwetting. It often causes psychological and social distress. Several contributing factors include:

Genetics - Children with a family history are at higher risk.

Bladder dysfunction - Overactive or underactive bladders can contribute.

Hormonal imbalances - Especially a deficiency in antidiuretic hormone (ADH), which leads to excessive nighttime urine production.

NE is classified as:

Primary NE: The child has never achieved nighttime dryness.

Secondary NE: The child had achieved dryness but started wetting again.

It can also be:

Mono-symptomatic (nighttime only)

Non-mono-symptomatic (includes daytime symptoms)

Current Treatments:

Behavioral: Bedwetting alarms, bladder training

Pharmacological: Desmopressin (synthetic ADH), oxybutynin

Psychological: Counseling and emotional support

Role of Telerehabilitation:

Telerehabilitation is a branch of telehealth offering remote rehabilitation services via communication technologies. Benefits include:

Useful where direct provider access is limited

Cost-effective and time-saving

Increases access to care in underserved or rural areas

Particularly valuable during public health emergencies (e.g., COVID-19)

Reduces waiting times for therapy

Study Aim:

To assess the effectiveness of telerehabilitation-specifically lifestyle and dietary advice delivered remotely-in reducing the frequency of bedwetting in children with primary NE.

Methodology:

Design:

Randomized Controlled Trial (RCT)

Participants:

Inclusion Criteria:

Children aged 5-10 years

Diagnosed with primary NE

Bedwetting occurs more than 4 nights per week

Exclusion Criteria:

Secondary NE due to neurological/musculoskeletal/congenital conditions

On pharmacological treatment for NE

Recruitment:

Online via social media

Parents filled out a screening form

Informed consent obtained from caregivers

Sample size calculated using G-Power software

Group Allocation:

Study Group: Received telerehabilitation (lifestyle + dietary advice)

Control Group: Did not receive any intervention

Intervention Details (Telerehabilitation):

Duration:

1 week of intervention, following a 1-week baseline, with 1-week post-treatment follow-up

Components:

Lifestyle and Motivational Counseling (based on Hjalmas et al., 2004):

Reassurance ("You WILL become dry!")

Regular voiding and fluid intake routines

Encourage calm bedtime routines

Educate parents and child about normal bladder function

Dietary Advice (based on Pietro Ferrara et al., 2015):

Recommended Foods: Vegetables, cereals, eggs, yogurt, fruits (pineapple, banana), fish

Avoid at Evening: Milk, cheese, salty foods

Avoid Completely: Chocolate, caffeine, carbonated drinks, citrus juices

Outcome Measures:

Reduction in Wet Nights (per ICCS classification):

Non-responder: <50% reduction

Partial responder: 50-99% reduction

Full responder: 100% dry nights

Pediatric Quality of Life: Measured pre- and post-treatment

Assessment Procedure:

Week 1: Baseline recording of wet nights

Week 2: Intervention period (study group only)

Week 3: Follow-up assessment for both groups

Data Collection & Analysis:

Demographics: Age, sex, weight, family history of NE

Clinical data: Frequency of wet nights

Descriptive stats: Means ± SEM for quantitative data; percentages for qualitative

Paired t-test: To compare outcomes before and after telerehabilitation

Expected Outcomes:

Reduction in bedwetting frequency in the study group receiving telerehabilitation

Improvement in quality of life metrics

Demonstrated feasibility and benefit of remote intervention in pediatric NE management

ELIGIBILITY:
Inclusion Criteria:

* Children aged 5 to 10 years.
* Diagnosed with primary nocturnal enuresis.
* Experience more than 4 wet nights per week.
* No prior pharmacological treatment for enuresis.
* Caregiver is willing to provide informed consent and participate in remote sessions.

Exclusion Criteria:

Diagnosis of secondary nocturnal enuresis due to:

* Neurological disorders
* Musculoskeletal problems
* Congenital abnormalities
* Currently receiving or recently received pharmacological treatment for nocturnal enuresis.
* Inability to participate in telehealth or remote intervention sessions.
* Caregiver does not consent to participation.

Ages: 5 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2025-06-29 (Actual); Primary Completion 2026-03-29 (Estimated); Study Completion 2026-03-29 (Estimated)

PRIMARY OUTCOMES:
number of wet nights/week | Baseline and 4 weeks after completion of telerehabilitation intervention
  The number of bedwetting episodes recorded by the caregiver during one week.
Pediatric Quality of Life scores | Baseline and 4 weeks after completion of telerehabilitation intervention
  Child and parent-reported outcomes using the Pediatric Quality of Life Inventory (PedsQL 4.0 Generic Core Scales). This validated tool measures physical, emotional, social, and school functioning. Total score ranges from 0 to 100, where higher scores indicate better quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of physical therapy kfs university, Kafr ash Shaykh, Kafr el-Sheikh Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Plan Description:
  The following specific Individual Participant Data (IPD) will be shared:
  Demographic Data:
  Participant age
  Sex
  Weight
  Family history of nocturnal enuresis (in parents or siblings)
  Clinical Baseline Data:
  Number of wet nights per week at baseline
  Type of enuresis (primary mono-symptomatic)
  Intervention Details:
  Group allocation (study vs. control)
  Telerehabilitation session logs (adherence to advice)
  Outcome Data:
  Number of wet nights post-intervention
  Classification according to ICCS criteria (non-responder, partial responder, responder)
  Pediatric quality of life scores (pre- and post-intervention)
  Adverse Events (if any):
  Reports of negative outcomes or non-compliance issues during the intervention
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: The individual participant data (IPD) and supporting documentation will be made available on Zenodo beginning 6 months after publication of the study results. The data will remain publicly accessible for a minimum of 5 years from the upload date.
Access Criteria: De-identified IPD, the study protocol, and data dictionary will be openly available to the public via Zenodo. Anyone may access and download the dataset under a Creative Commons license (e.g., CC BY 4.0). Users must agree to use the data for research or educational purposes only, with proper citation of the dataset and original publication.
URL: https://zenodo.org/